CLINICAL TRIAL: NCT03434886
Title: Evaluating Outcomes in European Cystic Fibrosis Patients With Access to Their Health Records: a Randomised Control Trial of a Registry Patient Portal
Brief Title: Outcomes in CF Patients Accessing Their Registry Health Records
Acronym: CFView
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cystic Fibrosis Registry of Ireland (Other)
Responsible Party: Principal Investigator, Abaigeal Jackson, Research Lead, Cystic Fibrosis Registry of Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CFView
Record Dates: First submitted 2018-02-08; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CF View (Experimental)
  Interventions: Other: CFView
- CF Educational videos (Active Comparator)
  Interventions: Other: CF educational videos
- CF View and videos (Active Comparator)
  Interventions: Other: CFView; Other: CF educational videos
- Usual standard of care (No Intervention)

INTERVENTIONS:
Other: CFView — Registry patient portal
  Arms: CF View; CF View and videos
Other: CF educational videos — CF educational videos
  Arms: CF Educational videos; CF View and videos

SUMMARY:
A multifactorial, parallel group, randomised control study in cystic fibrosis (CF) patients aged 13-30 years over an 18 month period. Patients will be offered read-only access to their CF registry electronic health record (CF View), or educational videos on CF (videos), or videos and CF View, or usual standard of care. The study aims are to examine the effect of patient access to C View on a range of clinical outcomes, health service usage, health literacy and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with CF
* registered with their national CF patient registry
* FEV1pp ≥40
* aged 13-30 years

Exclusion Criteria:

* organ transplantation
* FEV1pp <40

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 282 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
FEV1pp | 18 months
  forced expiratory volume in 1 second percentage predicted

SECONDARY OUTCOMES:
Health literacy | 12 months
  Health Literacy Survey - HLS- EU - Q16 score
Health-related quality of life | 12 months
  CFQr score - (Cystic Fibrosis questionnaire revised)
BMI | 18 months
  kg/m^2
Pulmonary exacerbations | 18 months
  pulmonary exacerbation requiring IV antibiotics
Hospitalisations | 18 months
  hospitalisation for treatment of pulmonary exacerbation

IPD SHARING:
Plan to Share IPD: No